Form Date: February 14, 2024



Department of Public Health Sciences 9201 University City Boulevard Charlotte, NC 28223-0001

## Consent to be Part of a Research Study

Title of the Project: Development and Implementation of a Self-Directed Violence Risk Assessment & Management Training Program for the North Carolina Department of Adult Corrections

Principal Investigator: Robert J. Cramer, Ph.D

University of North Carolina at Charlotte Co-investigator: Abigail Post, Ph.D. University of North Carolina at Charlotte Co-investigator: Sam Cacace, Ph.D. University of North Carolina at Charlotte Co-investigator: Jessamyn Moxie, Ph.D.

University of North Carolina at Charlotte Co-investigator: Ava Peters

NC Department of Adult Corrections Co-investigator: L. Jonathan Peiper, Ph.D. Study Sponsor: North Carolina Department of Health and Human Services

You are invited to participate in a research study. Participation in the training is mandatory per your position requirements at the North Carolina Department of Adult Corrections. However, <u>your participation in this survey research study is voluntary</u>. The following information is to help you decide whether or not to participate. If you have any questions, please ask.

#### **Important Information You Need to Know**

- The purpose of this study is to test and improve a pilot SDV risk assessment and management training program for correctional behavioral health clinicians. Participation in the training is mandatory per your position requirements at the North Carolina Department of Adult Corrections. However, your participation in this survey research study is voluntary.
- You will complete this required SDV risk assessment and management training program in-person at one of two sessions. The training will require eight (8) to twelve (12) hours of your time, and you will receive continuing education (CE) credits for the training.
- This training is being offered as standard CE training for NC DAC behavioral health clinicians and the NC-DAC has invited researchers from UNC Charlotte to assist in the development and assessment of the training content and its efficacy.
- No matter which training session you are assigned to, you will be asked to complete three (3) surveys: a baseline assessment survey and two follow-up assessment surveys (one-month after each training session). These surveys are optional, but will help us evaluate and improve the training.
- Each survey will take approximately 20-30 minutes to complete. The total time commitment for completing all three surveys is estimated to be 60-90 minutes. The training itself is estimated to take 8 hours; however all behavioral health clinicians are required to take the training. While your total time commitment is 9-9.5 hours, only 60-90 minutes are required for the optional surveys.
- The UNC Charlotte team will maintain a list of trainee email addresses linked to study-specific training IDs. Your email address will be used to enroll you in the training. The document linking your email address and study ID will be deleted once the training evaluation is completed.
- Dr. Peiper will not have access to your survey responses or whether you decide to participate in the optional research survey study. Choosing not to participate in the survey study portion of the training will not affect your job appraisal or performance review.
- You will be asked to enter your email address into each survey. This means your responses will be temporarily identifiable. The study team will use your email address to link survey responses. Email addresses will be deleted as soon as the data linkage process is completed, and your email address will be replaced with a random study ID number.

- Risks or discomforts from this research include infrequent emotional discomfort due to the sensitive nature of some questions, and rare social risk if you allow others to see your survey responses.
- There are no direct benefits to you by participating in the research survey study. There is no incentive for participation in the optional research survey administration. Choosing not to participate in this research will not affect the CE credit you will receive for participating in the training session. You will help us develop an evidence-based SDV prevention training that will improve care within NC DAC. We will also be able to spread the training program beyond North Carolina.

Please read this form and ask any questions you may have before you decide whether to participate in this survey research study.

## Why are we doing this study?

The purpose of this study is to test and improve a self-directed violence risk assessment and management training program for correctional behavioral health clinicians. Specifically, we are interested in gaining behavioral health clinician feedback to improve the training. We are also interested in how this training program impacts behavioral health clinician attitudes, knowledge, and risk assessment and management skills.

## Why are you being asked to be in this research study?

You are being asked to be in this study because you are over 18 years of age, live in the United States, and are currently employed as a North Carolina Department of Adult Corrections behavioral health clinician. Dr. Lewis Jonathan Peiper, PhD identified you as a person meeting these criteria.

## What will happen if I take part in this study?

You will only take part in one of the training sessions. If you choose to participate in this survey evaluation study, you will be asked to complete three voluntary surveys: at baseline, and follow-up 1 (one-month after the first group's training session) and follow-up 2 (one-month after the second group's training session). Survey items will address demographic information; training importance and intent; training feasibility and recommendations for improvement; and, SDV prevention knowledge, attitudes and practices. No Private Health Information (e.g., Social Security Number, address) is being requested. The time commitment for surveys will take approximately 60-90 minutes total to complete (20-30 minutes per survey). Dr. Peiper has indicated each behavioral health clinician will be provided release time over the study period to complete the training and voluntary surveys. (Dr. Peiper's authorization to use training time as work time will be in accordance with the agency's Training Leave Policy for mandatory or required training).

We will not collect any additional information.

# What benefits might I experience?

You will not directly benefit from being in this study, but you may gain insight into your own SDV prevention knowledge, attitudes, and skills. Also, others might benefit in that study results will inform the revision and sustainable implementation of the pilot SDV prevention training program.

#### What risks might I experience?

There is an infrequent chance you may experience mild emotional or psychological discomfort due to the sensitive nature of some questions. To minimize this risk, we have had the project reviewed by the Human Subjects Review Board and by experts in correctional SDV. If any question makes you uncomfortable, you may withdraw from research survey participation at anytime. If you feel any discomfort after having participated in this study there are a number of resources available to you.

- 1. Should you need assistance with your mental health, you can access the Employee Assistance Program (EAP) at (888) 298-3907 or (704) 717-5295 to speak with an experienced licensed counselor.
- 2. For non-emergent issues, you can access the S.H.I.E.L.D. program at 1-855-774-4353 (1-855-7SHIELD) for confidential peer support services.
- 3. You may also contact Dr. Peiper directly.
- 4. To locate psychological services beyond those offered by the NC DAC, you can access the American Psychological Association's Psychologist Locator (<a href="http://locator.apa.org">http://locator.apa.org</a>) to find a licensed counselor.

5. If you are experiencing any immediate distress, please call the National Suicide Prevention Lifeline at 988. You may also reach the national Crisis Text Line by texting HOME to 741741.

### **How will my information be protected?**

We plan to publish the results of this study. To protect your privacy, we will not include any information that could identify you. Data are confidential. You will be asked to enter your email address into each survey. This means your responses will be temporarily identifiable. The study team will use your email address to link survey responses. Email addresses will be deleted as soon as the data linkage process is completed, and your email address will be replaced with a random study ID number. Participant email addresses will be maintained in a secure, password protected DropBox folder (only study team members at UNC Charlotte will have password and file access). Dr. Peiper will not have access to survey responses, nor study IDs, in order to protect the privacy of your survey responses from your supervisor(s). Survey data will be downloaded in an anonymous group-level format stripped of identifiers (e.g., IP addresses). Once data analysis is complete, email addresses linked with study ID numbers will be deleted no less than one month after study completion.

#### How will my information be used after the study is over?

The data/information collected will not be used or distributed for future research studies even if identifiers are removed

### Will I receive an incentive for taking part in this study?

There is no incentive for participation in this study. Remember, the CE credits offered for participating in the training program will not be affected if you choose not to participate in this research study.

#### What other choices do I have if I don't take part in this study?

The training is required by NC DAC. However, you may elect not to complete the survey study and you may withdraw from the study at any time.

# What are my rights if I take part in this study?

It is up to you to decide to be in this research study. Participating in this survey study is voluntary. Even if you decide to be part of the study now, you may change your mind and stop at any time. You do not have to answer any questions you do not want to answer.

#### Who can answer my questions about this study and my rights as a participant?

For questions about this research, you may contact either the study lead investigator or NC Department of Adult Corrections lead:

Robert Cramer, Ph.D. Associate Professor of Public Health sciences UNC Charlotte rcramer4@charlotte.edu (704) 687-6022 L. Jonathan Peiper, Ph.D.
Director of Behavioral Health
NC Department of Adult Corrections
lewis.peiper@ncdps.gov
(984) 255-6072

If you have questions about your rights as a research participant, or wish to obtain more information, ask questions, or discuss any concerns about this study with someone other than the researcher(s), please contact the UNC Charlotte Office of Research Protections and Integrity at 704-687-1871 or <a href="mailto:uncc-irb@charlotte.edu">uncc-irb@charlotte.edu</a>.

#### **Consent to Participate**

Remember, you are required by Dr. Peiper and the North Carolina Department of Adult Corrections to complete your SDV prevention training. The optional survey portion of the study is marked at the beginning and end of the training program. By clicking "yes, I agree to participate" below, you are agreeing to participate in the optional survey research study. By selecting "yes, I agree to participate," you will be directed to the baseline survey via Qualtrics.

| Make sure you understand what the study is about before you sign. You can save a screenshot picture of this document for your records or request it from study investigators. If you have any questions about the study after you sign, you can contact the study team using the information provided above. |
|---|
| I understand what the study is about, and my questions so far have been answered. By clicking "yes, I agree to participate" in the optional research survey study portion of the training. |
| YES, I agree to participate |
| NO, I do not want to participate |